CLINICAL TRIAL: NCT06539091
Title: A Single-Arm, Open, Multicenter, Exploratory Clinical Study of Fluzoparib in Combination With Apatinib Mesylate for Maintenance Therapy in Stage III-IV Ovarian Cancer (FAT-1)
Brief Title: Fluzoparib in Combination With Apatinib Mesylate for Maintenance Therapy in Stage III-IV Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhou ying-FAT-1
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Epithelial Ovarian Cancer; Efficacy; Safety; Bone Mineral Density; Tolerability
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib group (Experimental): During the treatment period, subjects were given fluazoparib capsules orally, two capsules/dose (50mg/capsule) twice daily, taken orally in the morning and in the evening, as a continuous dosage. Treatment will continue until an event occurs that meets the criteria for discontinuation of treatment.
  Interventions: Drug: Fluzoparib
- Apatinib Mesylate group (Experimental): During the treatment period, subjects will also receive oral apatinib mesylate tablets, one tablet/dose (250 mg/tablet), once daily, continuously. Treatment will continue until an event occurs that meets the criteria for discontinuation of treatment.
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Fluzoparib — The study treatment was followed by a 3-week treatment cycle. First day of each dosing cycle, subjects are required to complete various examinations, including vital signs, physical examination, laboratory examination, physical status score, and BMD testing to evaluate the safety and tolerability of continued treatment.
  Arms: Fluzoparib group
Drug: Apatinib Mesylate — The study treatment was followed by a 3-week treatment cycle. First day of each dosing cycle, subjects are also required to complete various examinations, including vital signs, physical examination, laboratory examination, physical status score, and BMD testing to evaluate the safety and tolerability of continued treatment.
  Arms: Apatinib Mesylate group

SUMMARY:
This study is a single-arm, open, multicenter, exploratory clinical study to observe and evaluate the efficacy and safety of fluazoparib combined with apatinib mesylate in the treatment of patients with ovarian cancer.

Patients with epithelial ovarian, fallopian tube, and primary peritoneal cancers will be selected as the study population with Progression-Free Survival (PFS) as the primary study endpoint, and Overall Survival (OS), Duration Of Response (DOR), Quality of Life Score QoL, Chemotherapy-Free Interval (CFI), Progression-Free Survival 2 (PFS-2), CA125 response criteria by GCGI, to access the safety、Bone Mineral Density (BMD) changes and the tolerability of fluazoparib in combination with apatinib mesylate.

The study is planned to enroll 51 subjects, all of whom will receive study treatment after being signed informed and screened.

DETAILED DESCRIPTION:
During the treatment period, subjects were given fluazoparib capsules orally, two capsules/dose (50mg/capsule) twice daily, taken orally in the morning and in the evening, as a continuous dosage. Subjects will also receive oral apatinib mesylate tablets, one tablet/dose (250 mg/tablet), once daily, continuously. Treatment will continue until an event occurs that meets the criteria for discontinuation of treatment.

Safety evaluations will be performed on Day 1 of each 3-week treatment cycle (vital signs, physical examination, laboratory examination, physical status score and BMD testing); imaging evaluations and once CA125 test will be performed every 6 weeks for the first 24 weeks of dosing, and every 9 weeks thereafter to assess efficacy, and for 12 months or until an event occurs that meets the criteria for treatment discontinuation. Dose suspension or downward adjustment may be made during the study period based on the occurrence of adverse events in subjects.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS: 0-1;

  * Initially treated patients with histologically or cytologically confirmed high-grade plasma ovarian cancer (HGSOC), fallopian tube cancer, primary peritoneal cancer, or endometrioid carcinoma of the ovary with FIGO stage III-IV;

    * No prior maintenance therapy with PARP inhibitors; ④Final use of a combination chemotherapy regimen of bevacizumab, paclitaxel and carboplatin; ⑤Good function of major organs; ⑥Subjects voluntarily enrolled in this study, signed an informed consent form, had good compliance, and cooperated with follow-up visits; ⑦The modeled CA-125 ELIMination rate constant K (KELIM) ≥ 1.

Exclusion Criteria:

* Patients concurrently enrolled in other clinical trials;

  * Previous maintenance therapy with PARP inhibitors combined with anti-angiogenic drugs;

    * Previous history of allergic reaction, hypersensitivity reaction, intolerance to antibody-based drugs;

      * Previous significant allergy to drugs or food or other substances;

        * Subjects with untreated CNS metastases, previously treated with systemic, radical brain or meningeal metastases (radiotherapy or surgery), may be included if imaging confirms that stabilization has been maintained for at least 1 month and systemic hormone therapy (dose >10mg/day prednisone or other isotonic hormones) has been discontinued for >2 weeks without clinical evidence;

          * Those who are unable to swallow tablets normally, or have abnormal gastrointestinal function that, in the judgment of the investigator, may interfere with drug absorption;

            * Have experienced clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months prior to randomization, such as peptic bleeding, bleeding gastric ulcer or suffering from vasculitis, etc. If the fecal occult blood is positive at the baseline period, it can be reviewed, and if it is still positive after review, combined with the clinical judgment, and if necessary, gastroscopy can be performed; ⑧The presence of currently uncontrolled malignant pleural fluid, ascites or pericardial effusion (defined as not effectively controlled by diuretics or puncture, as judged by the investigator);

              * Presence of uncontrolled comorbidities including, but not limited to: active HBV or HCV infection, known HIV infection or history of AIDS, active syphilis, active tuberculosis, active infections, uncontrolled hypertension, symptomatic cardiac insufficiency, and active bleeding;

                * Previous (within 5 years) or concurrent other untreated malignant tumors, except for cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and breast cancer without recurrence > 3 years after completion of radical surgery; ⑪Women during pregnancy or lactation; ⑫Having taken a drug that clearly affects the study drug within 30 days or 5 half-lives (whichever is longer) prior to enrollment; ⑬In the judgment of the investigator, the subject has other factors that may cause this study to be forcibly terminated midway, such as other serious illnesses (including psychiatric illnesses) that require comorbid treatment, serious laboratory test abnormalities, accompanied by family or social factors that would affect the subject's safety, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 year
  Progression-Free Survival (PFS) is defined as the time interval between a patient's diagnosis of gynecological malignancy and the first occurrence of progression of the disease or death from any cause.

SECONDARY OUTCOMES:
OS | 2 year
  Overall Survival (OS) was defined as the time interval between a patient's diagnosis of gynecologic malignancy and death from any cause or the end of the last follow-up date.
DOR | 2 year
  Duration Of Response (DOR) is defined as the time from when a patient reaches first remission (including complete or partial remission) to when the disease re-progresses.
QoL | 2 year
  Quality of Life Score (QoL) is a score that assesses a patient's overall physical, psychological, social, and environmental well-being through a standardized questionnaire or scale.The scale has a full score of 60, with a very poor score of <20, a poor score of 21-30, a fair score of 31-40, a better score of 41-50, and a good score of 51-60.
PFS-2 | 2 year
  Progression-Free Survival 2 (PFS-2) defined as the time from patient randomization to completion of secondary therapy after disease re-progression or patient death.
AE | 2 year
  Adverse events (AE) are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)